CLINICAL TRIAL: NCT05129709
Title: Addressing Communication Challenges Confronting Older African Americans With Multiple Chronic Conditions and Their Family Caregivers
Brief Title: Black Health Identification Program (B-HIP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Deborah Ejem, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300007623; Kornfeld Scholar Award (Other Grant/Funding Number: National Palliative Care Research Center)
Record Dates: First submitted 2021-07-28; First posted 2021-11-22 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Multiple Chronic Conditions; Family Members
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: The Social Cognitive Theory (SCT) and the Health Belief Model (HBM) inform this proposal. The SCT posits that human behavior is determined by expectancies- of culture, potential outcomes, and self-efficacy- and incentives. The HBM holds that health-related behavior depends on motivation, the belief that one is susceptible to serious illness, and the belief that following provider advice will reduce the threat. Concepts of health beliefs, self-efficacy, and culture must be considered when developing effective interventions for value solicitations and behavior change. This is especially true for older AAs in the Deep South, who report different lived experiences and experiences with medical icare than Whites. Patient-centered care cannot be realized for AAs without reshaping interventions to consider factors important to seriously ill older AAs with MCCs. Reframing discussion in a culturally-responsive manner is necessary to establish patient and FCG preferences prior to a health crisis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "My Health Priorities" Identification Program (Experimental): The intervention, the "My Health Priorities" Identification Program consists of four self-directed, web-based modules intended to guide patients with MCCs in identifying their own health priorities. These priorities can then be used to guide discussions with family caregivers and clinicians regarding specific goals and preferences that they wish to guide future treatment decisions. Most models of palliative care have been developed based on white middle-class populations and may not apply to African Americans (AA) who have a very different cultural value set.
  Interventions: Behavioral: "My Health Priorities" Identification Program

INTERVENTIONS:
Behavioral: "My Health Priorities" Identification Program — The web-based "My Health Priorities" Identification Program may improve values solicitation and operationalization skills in primary care, but has not been optimized for AAs with MCCs and their FCGs. The Program is a facilitator-led evidence- and values-based care communication model for patients, clinicians, and caregivers that has reduced patient-reported treatment burden by aligning value-based priorities with treatment. The web-based program assists patients in identifying their health priorities as they complete t four online modules that help them to identify specific and actionable health goals and preferences. The final result can be printed and brought to the clinic or uploaded to the Electronic Medical Record to inform subsequent healthcare decision making. Unrecognized cultural preferences of AAs, including the important role of R/S beliefs and family-centered values, can interfere with adequate healthcare communication resulting in healthcare disparities and inequities.

SUMMARY:
Nearly 69% of African American (AA) Medicare beneficiaries have multiple chronic conditions (MCCs) such as cancer and cardiopulmonary diseases. Older age and MCCs are guideline-recommended indications for referral to early palliative care to assist with effective communication and value-solicitation surrounding treatment decision-making. Studies have shown that early palliative care participation achieves beneficial goals of care communication, quality of life (QOL), symptom burden, and mood in older adults with cancer and heart failure as well as among their family caregivers. However, older AAs with MCCs, especially those living in the Deep South, are less likely to have access to early palliative care, even though they generally experience higher symptom burden, healthcare use, and poorer communication around goals of care. This disparity in palliative care use may be, in part, to a lack of culturally-responsive care practices that effectively activate AAs with MCCs to identify their own values and priorities for end-of-life care. While efficacious communication models exist, few have been tested in culturally-diverse samples. Guided by the theory of Social Cognitive Theory and Health Behavior Model, this study's purpose is to conduct a formative evaluation of a Self-directed "My Health Priorities" Identification Program to determine cultural acceptability and feasibility of use in among AAs with MCCs in a primary care setting. The 2-phase study specific aims are to:

Aim 1. (Phase 1) Conduct a single-arm formative evaluation trial of Self-directed "My Health Priorities" Identification Program to determine acceptability and feasibility with a sample of 20 AA patients with MCCs and FCGs and adapt for future efficacy testing.

Aim 2. (Phase 2) To examine the ability of the dyads to complete pre- and post-test measures of perception of care, treatment burden, shared decision-making, and communication exchange.

The findings from the research will directly inform a small-scale pilot grant that will assess acceptability, feasibility, and potential efficacy of a values solicitation and operationalization intervention for AAs with MCCs and caregivers.

ELIGIBILITY:
Inclusion Criteria for Patients

* African American (AA)
* ≥ 65 years
* has at least two of the following chronic conditions: cancer, heart disease, kidney disease, liver disease
* English-speaking
* cognitively able to participate in decision-making discussions
* reliable internet and telephone access
* FCG willing to participate in study

Inclusion Criteria for FCG

* AA

  * 18 years
* identified by patient as his/her primary FCG
* English-speaking; and 5) reliable internet and telephone access.

Exclusion Criteria for Patients and FCG

* Axis I psychiatric disorder (schizophrenia, bipolar disorder), dementia
* active substance use disorder
* living in a nursing home or assisted living facility residence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
A single arm formative evaluation (qualitative interviews) exploring acceptability of the program | one-time interview six weeks following baseline questionnaires
  Semi-structured interview of patients with multiple chronic illness (MCC)
A single arm formative evaluation (qualitative interviews) exploring acceptability of program | one-time interview six weeks following baseline questionnaires
  Semi-structured interview of family caregivers (FCG) of patients with MCC
System Usability Scale (ISUS) | one-time interview six weeks following baseline questionnaires
  Measures usability of web-based applications and programs in both patients and FCG,. subscales evaluate how learnable and usable the tested program is; 10 items, 5 items are scored positively and 5 items are scored negatively using a 5 point likert scale with 5 indicating strongly agree and 1 indicating strongly disagree
Program Completion Statistics | one-time interview six weeks following baseline questionnaires
  Usability statistics will be obtained about the length of time the participant engaged with the program, and module completion rates
Older Patient Assessment of Chronic Illness Care (O-PACIC) | Baseline
  Questionnaire of perception of care among patients with MCC. The questionnaire consists of 10 items scored on a 5 point likert scale with 5 indicating "almost always" and 1 indicating "almost never". Higher scores thus reflect patients' perception of better care.
Treatment Burden Questionnaire (TBQ) | Baseline
  Patients with MCC perception of QOL and treatment burden related to chronic illness; 15 items rated on a ten point scale with 0 indicating that the item "is not a problem" and 10 indicating that the item reflects a "big problem".
Clinical Shared Decision Making Questionnaire (CollaboRATE) | Baseline
  Patients with MCC-reported measure of clinical shared decision-making; 3 items requiring open-ended responses (no scale)
Bakas Caregiver Outcomes (BCOS) | Baseline
  Measures FCG social function, subjective well-being, and somatic health; 10 items rated on a 7 point likert scale with -3 reflecting "changed for the worst" and +3 indicating "changed for the better".
Shared Care Instrument (SCI) | Baseline
  PT and FCG's perception of communication exchange regarding illness experience, subscales include communication, decision making, and reciprocity; 19 items divided into 3 summary scales, each item is scored in likert format from 0 to 5 with 0 indicating "completely disagree" and 5 indicating "completely agree". On the communication subscale a higher score indicates better communication. For the patient decision making subscale, higher scores indicate better patient decision making. For the patient reciprocity scale, higher scores indicate more reciprocity between patient and caregiver.
Change in Older Patient Assessment of Chronic Illness Care (O-PACIC) | 18 weeks post-baseline
  Measure of older patient perception of primary care delivery; 10 items scored on a 5 point likert scale with 1 indicating "almost never" and 5 indicating "almost always". Higher scores reflect that patients have a more positive feeling about their care.
Change in Treatment Burden Questionnaire (TBQ) | 18 weeks post-baseline
  Patients with MCC perception of QOL and treatment burden related to chronic illness; 15 items rated on a ten point scale with 0 indicating that the item "is not a problem" and 10 indicating that the item reflects a "big problem".
Change in Clinical Shared Decision Making Questionnaire (CollaboRATE) | 18 weeks post-baseline
  Patients with MCC-reported measure of clinical shared decision-making; 3 items requiring open-ended responses (no scale)
Change in Bakas Caregiver Outcomes (BCOS) | 18 weeks post-baseline
  Measures FCG social function, subjective well-being, and somatic health; 10 items rated on a 7 point likert scale with -3 reflecting "changed for the worst" and +3 indicating "changed for the better".
Change in Shared Care Instrument (SCI) | 18 weeks post-baseline
  PT perception of communication exchange regarding illness experience, subscales include communication, decision making, and reciprocity; 19 items divided into 3 summary scales, each item is scored in likert format from 0 to 5 with 0 indicating "completely disagree" and 5 indicating "completely agree". On the communication subscale a higher score indicates better communication. For the patient decision making subscale, higher scores indicate better patient decision making. For the patient reciprocity scale, higher scores indicate more reciprocity between patient and caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ejem, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Whitaker Clinic at the University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ejem D, Bakitas M, Durant RW, Parker TN, Oppong KD, Esterson J, Odom JN, Wells RD, Boockvar K, Tinetti ME. Exploring the Acceptability and Feasibility of a Self-directed Approach to Identifying Health Priorities in a Sample of Southern Older African American Adults with Multiple Chronic Conditions. J Racial Ethn Health Disparities. 2025 May 23. doi: 10.1007/s40615-025-02469-8. Online ahead of print. PMID 40410637